CLINICAL TRIAL: NCT07109089
Title: Heart Rate Vs. Race Pace-Based Prescription Training: Which Training Method Leads To Intended Execution In Recreational Distance Runners?
Brief Title: Heart Rate Vs. Race Pace-Based Prescription Training in Recreational Distance Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Arturo Casado, Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IND/22HUM-23661
Record Dates: First submitted 2025-07-07; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Exercise Response; Physical Fitness; Athletic Performance; Running Endurance
Keywords: Endurance prescription; HIIT; Recreational runners; Excercise monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Race Pace Group (Experimental): Participants follow a training program based on race pace zones, including both low-intensity sessions and high-intensity intervals.
  Interventions: Other: Race Pace-based training
- Heart Rate Group (Experimental): Participants follow a training program based on heart rate zones, including both low-intensity sessions and high-intensity intervals.
  Interventions: Other: Heart Rate-Based Training

INTERVENTIONS:
Other: Race Pace-based training — Participants complete one week of endurance training based on race pace zones individually determined from a 5-km time trial performance. The program includes both low-intensity continuous runs and high-intensity interval training sessions.
  Arms: Race Pace Group
Other: Heart Rate-Based Training — Participants complete one week of endurance training based on heart rate zones individually determined from ventilatory threshold assessments. The program includes both low-intensity continuous runs and high-intensity interval training sessions.
  Arms: Heart Rate Group

SUMMARY:
The goal of this randomized controlled trial is to compare adherence to training prescription-defined as the percentage of time spent within the prescribed intensity zone-using either a race pace-based method or a heart rate-based method in male and female recreational distance runners.

The main research questions are:

* Which training prescription method leads to greater adherence in recreational runners?
* Which method results in more accurate execution of low- and high-intensity interval training sessions?

Participants will undergo anthropometric and physiological assessments to determine training zones based on ventilatory thresholds. In addition, a 5-km time trial will be performed on a standard track to establish individual race pace zones.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female recreational endurance runners
* minimum of four training sessions per week
* at least three of consistent endurance training experience

Exclusion Criteria:

* current smokers
* diagnosed metabolic disorders
* any cardiovascular, pulmonary, or orthopedic condition that may interfere with exercise performance or safety

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Maximal Oxygen Uptake (VO₂max) | Baseline
  VO₂max (mL·kg-¹·min-¹) measured during an incremental treadmill test to volitional exhaustion. Respiratory gases are collected breath-by-breath using a calibrated metabolic cart. The highest 30-second average of VO₂ is taken as VO₂max.
Time in Zone - Low-Intensity Training | Week 1 and week 2
  Total time (in minutes and % of intended time in zone) spent within the prescribed low-intensity training zone during each session, as determined by either heart rate (below first ventilatory threshold) or race pace (based on individual 5-km performance). Training zones are predefined per method and monitored via GPS watches and heart rate monitors.
Time in Zone - High-Intensity Interval Training (HIIT) | Week 1 and week 2
  Total time (in minutes and % of intended time in zone) spent within the prescribed high-intensity training zone during interval sessions, based on either heart rate (above second ventilatory threshold) or race pace (percentage of 5-km race pace). Time in zone is extracted from GPS and HR data post-session

SECONDARY OUTCOMES:
Body weight (kg) and Body Mass Index (BMI kg/m²) | Baseline
  These variables will be assessed to monitor changes in general health status and body composition throughout the intervention.
  Weight and height will be measured using a calibrated bio-electrical impedance analyzer (Tanita MC-780), with an accuracy of ±0.1 kg. Participants will be assessed barefoot, wearing light clothing, after an overnight fast and after voiding. Weight will be recorded in kilograms (kg) and height in meters (m), and BMI will be subsequently calculated as weight divided by height squared (kg/m²).
  No additional outcome measures will be collected in this assessment session.
Ventilatory thresholds | Baseline
  Oxygen uptake (VO₂, mL·kg-¹·min-¹) at the first and second ventilatory thresholds measured during an incremental treadmill test. Ventilatory thresholds are determined using standard gas exchange methods (e.g., V-slope, ventilatory equivalents).

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Casado, PhD, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Cam. del Molino, 5, Fuenlabrada, Madrid, Fuenlabrada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranieri LE, Casado A, Martin D, Trujillo-Colmena D, Gil-Arias A, Kenneally M, Jimenez A. Performance and Physiological Effects of Race Pace-Based Versus Heart Rate Variability-Guided Training Prescription in Runners. Med Sci Sports Exerc. 2025 Jul 1;57(7):1510-1522. doi: 10.1249/MSS.0000000000003671. Epub 2025 Feb 12. PMID 39935030